CLINICAL TRIAL: NCT03599583
Title: Improving HPV Vaccination Delivery in Pediatric Primary Care: The STOP-HPV Trial 3. Comparison of Prompts (in the Presence of Communication Skills and Performance Feedback) and Standard of Care
Brief Title: The STOP-HPV Trial 3: Prompts Intervention
Acronym: STOP-HPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, Executive Vice-Chair and Vice-Chair for Research, Department of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3R01CA202261 (NIH); R01CA202261 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Immunization; Vaccination
Keywords: HPV; Vaccination; Practice based intervention

STUDY DESIGN:
Intervention Model Description: RCT study design will test the impact of the prompts intervention to reduce missed opportunities and raise HPV vaccine rates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Arm 1 will receive the STOP-HPV prompts intervention
  Interventions: Behavioral: STOP-HPV prompts intervention
- Control (No Intervention): Arm 2 will receive standard of care

INTERVENTIONS:
Behavioral: STOP-HPV prompts intervention — This intervention will be the addition of the prompts intervention (in the presence of communication skills training and continued performance feedback).
  Arms: Intervention

SUMMARY:
Most adolescents who receive human papillomavirus (HPV) vaccine are vaccinated in pediatric practices, yet missed opportunities (MOs) for HPV vaccination occur often and lead to low HPV vaccination rates. This study is part of a series of cluster randomized clinical trials (RCTs) that will test the effectiveness (and cost-effectiveness) of the addition of prompts (period 3) to performance feedback (period 2, continued through period 3) and training providers previously received on HPV vaccine communication (period 1) to reduce MOs and increase HPV vaccination rates.

DETAILED DESCRIPTION:
This intervention will incorporate prompts via electronic health record (EHR) (e.g. alerts in electronic charts indicating patient is due for vaccination) and study practice staff prompts (reminders from study staff that a patient is due for vaccination, e.g. placing Vaccine Information Statements (VISs) on desk) to study practitioners that encourage HPV vaccination at all visits. An initial learning module on practitioner prompts will highlight how study practices can consistently implement both EHR and staff HPV vaccination prompts at all visits. Throughout the intervention, text message mini-lessons will remind participants how to best use prompts via EHR and/or office staff to improve HPV vaccination rates. This trial focuses on study period 3 where study periods are as follows:

Period 0: Baseline period, prior to the randomization of practices into intervention arms

Period 1: Arm-1 intervention study practices receive communication skills training; Arm-2 comparison study practices provide standard of care. Period 2: Arm-1 intervention study practices add performance feedback, building upon their prior training in communication skills; Arm-2 comparison study practices continue delivering standard of care. Period 3: Arm-1 intervention study practices add prompts, building upon prior communication skills and performance feedback; Arm-2 comparison study practices continue with standard of care.

Due to the COVID-19 pandemic, an additional 15-month study period (Pause Period) was introduced between feedback (Period 2) and prompts (Period 3). No study activities were undertaken during this time.

The prompts intervention effect will be interpreted within the context of the previous periods (Periods 0, 1 and 2) and the pause period.

ELIGIBILITY:
Practice Inclusion Criteria:

* The practice provides HPV vaccination services to adolescents.
* The practice is part of Physician's Computer Company (PCC), Office Practicum (OP) or (a) yet-to-be selected health system(s).
* The practice has had the same EHR system in place for a year or more (with special consideration on a case by case basis if they are close to but not do not reach a year).
* The practice agrees to not participate in other HPV-related QI projects or research interventions during the study period (with special consideration on a case by case basis).

Practice Exclusion Criteria:

* The practice plans to change EHR systems in the next three years.
* The practice participated in the last year, is currently engaged in, or plans to participate in an office-based HPV-related quality improvement (QI) project or research intervention during the study period (with special consideration on a case by case basis).
* Estimated 20% or more of adolescents at the practice receive HPV vaccinations at schools or health department clinics (given standard practice and published data, the investigators expect that few to no practices will need to be excluded based on this restriction).

Patient inclusion criteria:

-All patients of participating practices (intervention and comparison) aged 11-17 years who have at least 1 visit to the practice within the past two years.

Patient exclusion criteria:

-None apart from age of patients (above).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of missed vaccination opportunities among all clinicians | The 12-month portion of the pause period immediately preceding initiation of prompts and the 6-month prompts period, excluding the 4-week ramp-up.
  Change in the rate of missed vaccination opportunities separately by dose (initial vs. subsequent) and visit type (preventive vs. acute) among all clinicians.
Change in the rate of missed vaccination opportunities among consenting clinicians | The 12-month portion of the pause period immediately preceding initiation of prompts and the 6-month prompts period, excluding the 4-week ramp-up.
  Change in the rate of missed vaccination opportunities separately by dose (initial vs. subsequent) and visit type (preventive vs. acute) among consenting clinicians

SECONDARY OUTCOMES:
Change in the rate of missed vaccination opportunities among clinicians, excluding practices that failed to meet inclusion criteria throughout the study period. | The 12-month portion of the pause period immediately preceding initiation of prompts and the 6-month prompts period, excluding the 4-week ramp-up
  Change in the rate of missed vaccination opportunities separately by dose (initial vs. subsequent) and visit type (preventive vs. acute) excluding practices that failed to meet inclusion criteria throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: No